CLINICAL TRIAL: NCT06938750
Title: A Pilot Study of a Novel Medical Device for Pharmacological Therapy: The SecHold Device
Brief Title: Novel Medical Device for Pharmacological Therapy
Acronym: Sechold
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SecHold Baby
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Vascular Access; Vascular Access Complication; Vascular Access Complications; Catheter Malfunction; Catheter Infection; Therapeutic Drug Management; Nurse; Nurse Based Care Management; Innovative Procedures
Keywords: VASCULAR ACCESS; CATHETER; THERAPY; COMPLICATION; DEVICE; CENTRAL VASCULAR ACCESS

STUDY DESIGN:
Intervention Model Description: A clinical trial was carried out in an intensive care unit of the University Hospital of Navarra, a tertiary hospital reference center in intensive care in Navarra, in the north of Spain; where the use and clinical validation process of a newly created device registered by European patent as a utility model was implemented. This study was made over a period of 6 months, from June 2021 to December of the same year; after internal authorization from the center where the clinical validation process has been carried out and from the local ethics committee (pyto2019/47).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL (No Intervention): FIXATION OF VASCULAR ACCESSES WITH INFUSION OF THERAPY MAINTAINED IN THE TRADITIONAL WAY, DIRECTLY TO A THREE-WAY TAP AND EXTENSION FOR CONNECTION TO A CENTRAL DEVICE.
- INTERVENTION (Experimental): FIXATION OF VASCULAR ACCESSES WITH INFUSION OF THERAPY MAINTAINED IN THE TRADITIONAL WAY, DIRECTLY TO THREE-WAY TAP AND EXTENSION FOR CONNECTION TO CENTRAL DEVICE INCORPORATING THE SECHOLD GRIP SYSTEM FOR ATTACHMENT OF MULTIPLE DROPPERS TO IT, WITH LABELING AND ATTACHMENT TO BED/CRADLE, DROPPER STICK OR PATIENT/CARRIER CLOTHING.
  Interventions: Device: SECHOLD DEVICE

INTERVENTIONS:
Device: SECHOLD DEVICE — PLACEMENT OF A MULTIPLE THERAPY GRIPPING DEVICE TO FIX THE DRIPPER SYSTEMS ALONG ITS PATH TO SOME SURFACE OR SPACE, AVOIDING IT TO REMAIN IN THE AIR, WITHOUT MARKING OR LABELING AND FAVORING ITS ORGANIZATION. SECHOLD is a vascular access fixation device designed for critical clinical environments such as ICU and operating rooms. It allows the simultaneous connection of 3-6 parenteral therapies to the same vascular access, ensuring clear and protocolized identification of each drug by means of labels with name, concentration and infusion range, in addition to a universal color code. This reduces the risk of drug administration errors and facilitates optimal visualization of essential information. SECHOLD also organizes infusion systems connected to the same vascular access, preventing knots and pulls that can compromise catheter integrity in case of accidental infusion bag drops.
  Arms: INTERVENTION

SUMMARY:
Background: Different co-creation methods were used to design and prototype a new fixative device for multiple intravenous therapies with the ability to control and identify the pharmacological therapy administered to a patient. Objectives: To validate a newly created device for the reduction of complications related to the use of intravenous therapy Methods: A multidisciplinary team composed of eight professionals specializing in the field of critical care and an engineering professional in industrial design was responsible for collecting, evaluating, and materializing the ideas and needs arising from clinical practice in a device that met the standards of the same.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the intensive care unit
* patients with authorization to take part in the study

Exclusion Criteria:

* Patients with pre-existing medical conditions: Patients with diseases affecting coagulation, such as hemophilia or thrombocytopathies, could be excluded.
* Active infection patients: Any patient with vascular access site infections or systemic infections may be excluded to avoid complications.
* Inability to give informed consent: Patients who are unable to understand or consent to participate in the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
To reduce the risk of complications associated with the number of pharmacological errors. | day 1, day 7, day 14, at 6 months after placement and start of the study
  Recognize the number of pharmacological errors (DRUG INTERACTION, WRONG DRUG, WRONG DOSAGE, WRONG SPEED) that have occurred
To reduce complications associated with accidental catheter withdrawals. | day 1, day 7, day 14, at 6 months after placement and start of the study
  Number of complications associated with accidental catheter withdrawals during the study period

SECONDARY OUTCOMES:
Reduce complications associated with venous catheter placement and maintenance (thrombosis, phlebitis, catheter obstruction). | day 1, day 7, day 14, at 6 months after placement and start of the study
  Number of complications associated with venous catheter placement and maintenance (thrombosis, phlebitis, catheter obstruction)

OTHER OUTCOMES:
Improved satisfaction of healthcare professionals operating the device. | day 1, day 7, day 14, at 6 months after placement and start of the study
  Satisfaction Questionnaire:
  A form used in the workplace with an overall satisfaction level will be used with a Liker scale of 1-10, with 1 being not at all satisfactory and 10 being maximum satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Marta M Ferraz-Torres, PHD, Principal Investigator — Fundación Miguel Servet
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No